CLINICAL TRIAL: NCT03831022
Title: Contribution of Capillary Refilling Time and Skin Mottling Score to Predict Intensive Care Unit Admission of Patients With Septic or Haemorrhagic Shock Admitted to the Emergency Department
Brief Title: Usefulness of Capillary Refill Time and Skin Mottling Score to Predict Intensive Care Unit Admission
Acronym: TRCMARBSAU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hôpital Necker-Enfants Malades (Other)
Collaborators: Hôpital Cochin (Other); University Grenoble Alps (Other); University Hospital, Strasbourg, France (Other); Poitiers University Hospital (Other); Begin Military Hospital (Unknown); Argenteuil Hospital (Unknown); University Hospital, Limoges (Other); University Hospital, Marseille (Other)
Responsible Party: Principal Investigator, Romain Jouffroy, MD, Hôpital Necker-Enfants Malades
Other Study IDs: 2018-A02588-47
Record Dates: First submitted 2019-02-03; First posted 2019-02-05 (Actual); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Shock, Septic; Shock, Hemorrhagic
Keywords: shock; sepsis; haemoragy; intensive care unit; prediction
MeSH Terms: conditions — Shock, Septic; Shock, Hemorrhagic; Shock; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Capillary refill time and skin mottling score measurement at the admission to the emergency department — Patients who meet the inclusion criteria and none of the non-inclusion criteria will benefit from capillary refill time and skin mottling score measurement at the admission to the emergency department (ED) and followed during their hospital stay to precise the destination after ED (home, ICU, ward) and 30- and 90-days mortality after hospital admission.

SUMMARY:
In the emergency department (ED), the severity assessment of shock is a fundamental step prior to the admission in intensive care unit (ICU). As biomarkers are time consuming to evaluate severity of the micro and macro-circulation alteration, capillary refill time and skin mottling score are 2 simples, available clinical criteria validated to predict mortality in the ICU.

The aim of this study is to provide clinical evidence that capillary refill time and skin mottling score assessed in the ED also predict ICU admission of patients with septic or haemorrhagic shock.

DETAILED DESCRIPTION:
This trial is an observational, non-randomized controlled study. A total of 1500 patients admitted to the ED for a septic or hemorrhagic shock will be followed.

The primary outcome is the admission to the ICU.

The study will not impact the treatments provided to each patient. Capillary refill time and skin mottling score will not be taken into account to decide patient's treatments and/or ICU admission. Patients will be followed during their hospital stay in order to precise their destination after ED (home, ICU, ward) and 28- and 90-days mortality after hospital admission.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Skin mottling score> 2 and/or capillary refill time > 3secondes associated with at least one of the followings measured at the ED admission by the nurse in charge of the patient:

   1. Systolic blood pressure < 90mmHg or blood pressure decrease of 30% at least for patients with high blood pressure history
   2. Heart rate > 120 beats per minute
   3. Respiratory rate > 22 movements per minute
   4. Glasgow coma scale < 13.

Exclusion Criteria:

1. Age < 18 years
2. Pregnancy
3. Serious co morbid conditions with a not to be reanimated status known at the ED admission
4. Patients with guardianship or curator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to the ED for septic or haemorrhagic shock
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2018-12-17 (Actual); Primary Completion 2020-12-17 (Estimated); Study Completion 2020-12-17 (Estimated)

PRIMARY OUTCOMES:
Rate of ICU admission after ED. | 2 days
  The rate of ICU admission after ED will be monitored for each patient

SECONDARY OUTCOMES:
Mortality on day 30 after hospital admission | 30 days
  The vital status (alive or deceased) will be recorded on day 30 after hospital admission
Mortality on day 90 after hospital admission | 90 days
  The vital status (alive or deceased) will be recorded on day 90 after hospital admission

CONTACTS AND LOCATIONS:
Locations (1):
- Necker enfants malades Hospital, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pottecher T, Calvat S, Dupont H, Durand-Gasselin J, Gerbeaux P; SFAR/SRLF workgroup. Haemodynamic management of severe sepsis: recommendations of the French Intensive Care Societies (SFAR/SRLF) Consensus Conference, 13 October 2005, Paris, France. Crit Care. 2006;10(4):311. doi: 10.1186/cc4965. PMID 16941754
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Background] Pickard A, Karlen W, Ansermino JM. Capillary refill time: is it still a useful clinical sign? Anesth Analg. 2011 Jul;113(1):120-3. doi: 10.1213/ANE.0b013e31821569f9. Epub 2011 Apr 25. PMID 21519051
- [Background] Ait-Oufella H, Bige N, Boelle PY, Pichereau C, Alves M, Bertinchamp R, Baudel JL, Galbois A, Maury E, Guidet B. Capillary refill time exploration during septic shock. Intensive Care Med. 2014 Jul;40(7):958-64. doi: 10.1007/s00134-014-3326-4. Epub 2014 May 9. PMID 24811942
- [Background] Ait-Oufella H, Lemoinne S, Boelle PY, Galbois A, Baudel JL, Lemant J, Joffre J, Margetis D, Guidet B, Maury E, Offenstadt G. Mottling score predicts survival in septic shock. Intensive Care Med. 2011 May;37(5):801-7. doi: 10.1007/s00134-011-2163-y. Epub 2011 Mar 4. PMID 21373821
- [Background] Lima A, Jansen TC, van Bommel J, Ince C, Bakker J. The prognostic value of the subjective assessment of peripheral perfusion in critically ill patients. Crit Care Med. 2009 Mar;37(3):934-8. doi: 10.1097/CCM.0b013e31819869db. PMID 19237899
- [Background] Lara B, Enberg L, Ortega M, Leon P, Kripper C, Aguilera P, Kattan E, Castro R, Bakker J, Hernandez G. Capillary refill time during fluid resuscitation in patients with sepsis-related hyperlactatemia at the emergency department is related to mortality. PLoS One. 2017 Nov 27;12(11):e0188548. doi: 10.1371/journal.pone.0188548. eCollection 2017. PMID 29176794
- [Background] Mrgan M, Rytter D, Brabrand M. Capillary refill time is a predictor of short-term mortality for adult patients admitted to a medical department: an observational cohort study. Emerg Med J. 2014 Dec;31(12):954-8. doi: 10.1136/emermed-2013-202925. Epub 2013 Sep 17. PMID 24045049
- [Background] Jouffroy R, Saade A, Tourtier JP, Gueye P, Bloch-Laine E, Ecollan P, Carli P, Vivien B. Skin mottling score and capillary refill time to assess mortality of septic shock since pre-hospital setting. Am J Emerg Med. 2019 Apr;37(4):664-671. doi: 10.1016/j.ajem.2018.07.010. Epub 2018 Jul 6. PMID 30001815